CLINICAL TRIAL: NCT00151008
Title: Investigator-Initiated, Double Blind, Vehicle-Controlled, Bilateral Comparison Trial of Bexarotene (Targretin) Gel 1% vs. Vehicle Gel in Combination With Narrow Band UVB Phototherapy for Moderate to Severe Psoriasis Vulgaris
Brief Title: Bexarotene With Narrow-Band UVB for Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Ligand Pharmaceuticals (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4405
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Psoriasis
Keywords: psoriasis; bexarotene; narrow band; UVB
MeSH Terms: conditions — Psoriasis | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bexarotene/NBUVB vs placebo NBUVB

SUMMARY:
To determine if bexarotene gel with NBUVB phototherapy is more effective than placebo plus NBUVB for moderate to severe plaque-type psoriasis.

DETAILED DESCRIPTION:
Subjects will be applying active gel or placebo to target lesions to each side of the body in a blinded manner. They will start at three times a week and increase to daily or even twice a day regimen if tolerated. After 2 weeks of application, NBUVB will be added to treatment regimen (whole body, three times a week). Total study time is 10 weeks.

ELIGIBILITY:
Inclusion Criteria

* Patient must be a male or female aged 18 years or older
* Patient must have moderate to severe psoriasis vulgaris of at least 3% body surface area involvement
* Patient must have failed prior topical therapy
* Patient must be willing to minimize sun exposure, to use sun blockers if deemed necessary by the Investigator and to avoid use of tanning booths or other ultraviolet (UV) light sources
* Women of childbearing potential must have a negative urine ß-HCG pregnancy test with a sensitivity of at least 50 mIU/mL within seven days prior to starting of study gels and repeated every four weeks while patient remains on the study gels. All females of childbearing potential must agree to use 2 effective contraceptive methods or remain sexually abstinent one month prior to initiation of study drug, during the entire study period, and for one month after the last application of Targretin® gel 1%. Acceptable methods of birth control include: condoms with spermicide; diaphragm with spermicide; cervical cap with spermicide; spermicidal sponge; intrauterine device (IUD), oral contraceptives, Depo-Provera; contraceptive implants; vasectomy; or abstinence.
* Male patients must agree to use condoms with sexual partners of childbearing potential during the entire period of treatment and for at least one month after treatment is discontinued.
* Patients who are not sexually active and are not using contraception, must agree to use an approved method of contraception (as described above) should they become sexually active during the study

Exclusion Criteria

* Failure to understand the consent form
* Inability to comply with protocol requirements
* Pregnancy
* Inadequate birth control method
* Lactation
* Contraindication to use of topical retinoids
* Concomitant psoriasis therapies except for emollients and OTC shampoos
* Systemic psoriasis therapies, systemic Vitamin A in doses > 15,000IU/day, PUVA, (psoralen plus ultraviolet A irradiation), UVB, topical psoriasis therapies (other than emollients and OTC shampoos), other retinoid class drugs or investigational drugs within the past 1 month
* Current skin cancer
* History of previous melanoma
* History of skin sensitizing diseases (such as SLE)
* Concurrent medical illness that would make participation in this clinical trial ill-advised
* Patient unwilling or unable to avoid prolonged exposure to the sun or other UV light sources

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2003-11; Study Completion 2005-08

PRIMARY OUTCOMES:
Mean decrease in target lesion size for drug- and placebo-treated sides. The mean and median changes in target lesion scores will be compared for drug- and vehicle-treated sides. Additionally, target lesions will be photographed.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Magliocco, MD, Principal Investigator — Rutgers, The State University of New Jersey